CLINICAL TRIAL: NCT01702051
Title: Autologous Pancreatic Islet Cell Transplantation for Improved Glycaemic Control After Pancreatectomy: Observational Study
Brief Title: Extending Indication for Islet Autotransplantation in Pancreatic Surgery
Acronym: AutoTx
Status: Recruiting | Type: Observational
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Lorenzo Piemonti, Director Islet Transplantation Program, Scientific Institute San Raffaele
Other Study IDs: 43-09/02/2012
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Diabetes
Keywords: Pancreatogenic diabetes; Autologou Islet Transplantation; Pancreas; Pancreatectomy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum, PBMC
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: patients with chronic pancreatitis treated with total or subtotal pancreatectomy
- 2: patients underwent completion pancreatectomy because of anastomotic leak after partial pancreatectomy
- 3: patients underwent pancreatoduodenectomy in which pancreatic anastomosis was made impracticable by technical difficulties and/or high risk of leakage
- 4: patients underwent extensive distal pancreatectomy for pancreatic lesions located at the neck

SUMMARY:
Islet autotransplantation (IAT) is a therapeutic approach used to prevent pancreatogenic diabetes or to reduce the severity of diabetes after a major pancreatectomy. Total pancreatectomy with IAT is being used almost exclusively for treatment of chronic pancreatitis. More recently, indications other than chronic pancreatitis have been reported including IAT after extended pancreatectomy performed for the resection of benign tumors of the mid-segment of the pancreas or IAT after total pancreatectomy for severe abdominal trauma In this study, we study our experience with IAT for the treatment of a broader population of patients undergoing pancreatic surgery including subjects with technically unfeasible or high risk pancreatic anastomosis during partial pancreatectomy and subjects undergoing completion pancreatectomy because of anastomosis leakage after pancreatoduodenectomy for nonmalignant or malignant diseases.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age

  * ability to provide written informed consent
  * fasting glycaemia <126 mg/dl without glucose-lowering medications.

Exclusion Criteria:

* Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the trial
* Diagnosis of intraductal papillary mucinous cancer, unless the absence of multifocal lesion is demonstrated by endoscopic US
* Presence of multifocal or residual disease at the pancreatic margin. If a malignat disease is the reason for the surgery, 1 cm of the pancreatic remnant in proximity to the pancreatic margin will be resected and sent for immediate pathologic analysis to confirm margin negativity and to rule out multifocal tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent partial or total pancreatectomy
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-02; Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Beta cell function | month 1, 3, 6, 12 and every year up to death
  Beta-cell function will be assessed by fasting C peptide, HbA1c,glycaemia, change in average daily insulin requirements, basal (fasting) and -10 to 120 min time course of glucose, C-peptide and insulin derived from the arginine test, beta-score and Transplant Estimated Function

SECONDARY OUTCOMES:
Incidence of complications after pancreatic surgery | 90 days from discharge
  Complications will be defined and graded according to the Novel Grading System classification ( DeOliveira et al 2006). A special emphasis is given to life-threatening and permanently disabling complications.

OTHER OUTCOMES:
Incidence of each individual postoperative complication | 90 days from discharge
  1. death
  2. pancreatic fistula defined according to the International Study Group on Pancreatic Fistula (Bassi C et al 2005)
  3. delayed gastric emptying (DGE) defined according to the International Study Group on Pancreatic Fistula (Wente et al 2007)
  4. intra-abdominal complications
  5. medical complications

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Piemonti, MD, Principal Investigator — Scientific Institute San Raffaele; Gianpaolo Balzano, MD, Study Director — Scientific Institute San Raffaele
Locations (1):
- Ospedale San Raffaele (OSR), Milan, Italy

REFERENCES:
- [Background] Balzano G, Piemonti L. Autologous islet transplantation in patients requiring pancreatectomy for neoplasm. Curr Diab Rep. 2014 Aug;14(8):512. doi: 10.1007/s11892-014-0512-2. PMID 24915889
- [Result] Balzano G, Maffi P, Nano R, Mercalli A, Melzi R, Aleotti F, Zerbi A, De Cobelli F, Gavazzi F, Magistretti P, Scavini M, Peccatori J, Secchi A, Ciceri F, Del Maschio A, Falconi M, Piemonti L. Autologous Islet Transplantation in Patients Requiring Pancreatectomy: A Broader Spectrum of Indications Beyond Chronic Pancreatitis. Am J Transplant. 2016 Jun;16(6):1812-26. doi: 10.1111/ajt.13656. Epub 2016 Mar 1. PMID 26695701
- [Result] Balzano G, Maffi P, Nano R, Zerbi A, Venturini M, Melzi R, Mercalli A, Magistretti P, Scavini M, Castoldi R, Carvello M, Braga M, Del Maschio A, Secchi A, Staudacher C, Piemonti L. Extending indications for islet autotransplantation in pancreatic surgery. Ann Surg. 2013 Aug;258(2):210-8. doi: 10.1097/SLA.0b013e31829c790d. PMID 23751451
- [Result] Balzano G, Maffi P, Nano R, Mercalli A, Melzi R, Aleotti F, De Cobelli F, Magistretti P, Scavini M, Secchi A, Falconi M, Piemonti L. Diabetes-free survival after extended distal pancreatectomy and islet auto transplantation for benign or borderline/malignant lesions of the pancreas. Am J Transplant. 2019 Mar;19(3):920-928. doi: 10.1111/ajt.15219. Epub 2019 Jan 23. PMID 30549450
- [Result] Balzano G, Nano R, Maffi P, Mercalli A, Melzi R, Aleotti F, Gavazzi F, Berra C, De Cobelli F, Venturini M, Magistretti P, Scavini M, Capretti G, Del Maschio A, Secchi A, Zerbi A, Falconi M, Piemonti L. Salvage Islet Auto Transplantation After Relaparatomy. Transplantation. 2017 Oct;101(10):2492-2500. doi: 10.1097/TP.0000000000001750. PMID 28358727
- [Result] Venturini M, Sallemi C, Colantoni C, Agostini G, Balzano G, Esposito A, Secchi A, De Cobelli F, Falconi M, Piemonti L, Maffi P, Del Maschio A. Single-centre experience of extending indications for percutaneous intraportal islet autotransplantation (PIPIAT) after pancreatic surgery to prevent diabetes: feasibility, radiological aspects, complications and clinical outcome. Br J Radiol. 2016 Aug;89(1064):20160246. doi: 10.1259/bjr.20160246. Epub 2016 Jun 21. PMID 27327404